CLINICAL TRIAL: NCT06825117
Title: Impact of Probiotic Supplementation on Urinary Tract Infections and Clinically Relevant Outcomes of Kidney Transplant Recipients
Brief Title: PRObiotics for KIdney Transplantation
Acronym: ProKiT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Udine, Italy (Other)
Collaborators: Winclove Probiotics B.V. (Industry); Institut AllergoSan (Unknown)
Responsible Party: Principal Investigator, Umberto Baccarani, Prof, MD PhD FEBS, University Hospital, Udine, Italy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 64/2024
Record Dates: First submitted 2024-10-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Urinary Tract Infections; Kidney Transplant Rejection; Kidney Transplant Infection; Dysbiosis
MeSH Terms: conditions — Urinary Tract Infections; Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group (Experimental)
  Interventions: Dietary Supplement: OMNi-BiOTiC® 41167
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: OMNi-BiOTiC® 41167 — The probiotic OMNi-BiOTiC® 41167 consists of 3g of 3 x 10^9 CFU total L. gasseri W15, L. plantarum W1, L. plantarum W21, B. lactis W51, L. acidophilus W70 and L. reuteri W192 per sachet of which two are to be taken each day. Additional non-probiotic components are cranberry-extract (0.01g), D-mannose (0,4 g), vitamin D (2,25µg), maize starch and hydrolyzed rice protein. All the strains in OMNi-BiOTiC® 41167 are specifically tested and selected for their inhibition potential against the known most common uropathogens like the uropathogenic Escherichia coli (UPEC), Klebsiella pneumonia, Proteus mirabilis and Entercoccus faecalis.
  Arms: Probiotic group
Dietary Supplement: Placebo — The placebo consists of all components of OMNi-BiOTiC® 41167, except the probiotic bacteria, cranberry-extract, D-mannose and vitamin D. It has the same smell, taste and texture as the OMNi-BiOTiC® 41167.
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to assess if dietary supplememtation with OMNi-BiOTiC® 41167 reduces the risk of urinary tract infections in kidney transplant recipients. It will also assess whether it reduces the risk of graft rejection, modify immunosuppressive regimen, improves post-transplant gastrointestinal and bladder microbiome, gastrointestinal symptoms and quality of life.

The main questions it aims to answer are:

* Does daily intake of OMNi-BiOTiC® 41167 reduce the incidence and number of episodes of urinary tract infections?
* Does daily intake of OMNi-BiOTiC® 41167 reduce the incidence and number of episodes of acute graft rejection?
* Does dietary supplementation with OMNi-BiOTiC® 41167 modify gut and bladder microbiome?
* Does dietary supplementation with OMNi-BiOTiC® 41167 modify tacrolimus metabolism and immunosuppressive state?
* Does dietary supplementation with OMNi-BiOTiC® 41167 improves gastrointestinal symptoms and quality of life? Researchers will compare drug OMNi-BiOTiC® 41167 to a placebo (a look-alike substance that contains no drug) to see if OMNi-BiOTiC® 41167 exerts any clinically relevant beneficial effect.

Participants will:

* Take OMNi-BiOTiC® 41167 or a placebo every day for 6 months
* Undergo clinical surveillance with seriated visit the clinics for checkups and laboratory analysis
* Provide seriated urine and stool samples for microbiome analysis
* Respond to seriated questionnaire on gastrointestinal symptoms and quality of life

DETAILED DESCRIPTION:
Background

Urinary tract infections (UTI) and graft rejection in kidney transplanted (KT) patients are currently the most frequent complications in the short-term, with a reported incidence of 17-51% and 6- 11% within the first year, respectively. The pathogenesis of such complications is tightly related and is determined by multifactorial mechanisms. Recent studies have shown that gut microbiota may have a crucial role in the pathogenesis of both post-KT UTI and graft rejection. Following transplantation, KT recipients show measurable alterations in microbial diversity, composition and function, and such gut dysbiosis may not only favor the proliferation of pathogens but also modify the immuno-inflammatory profile of recipients, inducing a pro- inflammatory state. Moreover, gut microbiota does metabolize immunosuppressant drugs, variably modifying their pharmacokinetic characteristics. A significant correlation between gut microbiota species and urine microbial isolates in a context of UTI have been consistently identified, and certain microbiota profiles have been alternatively associated with graft immune tolerance and graft rejection episodes. According to the International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statements, probiotics are defined as live microorganisms that, when administered in adequate amounts, confer a health benefit on the host.

Recent studies have shown that probiotic supplementation in KT recipients may variably improve kidney function in patients with chronic kidney disease as well as induce graft tolerance and decrease the risk of recurrent Clostridioides difficile infection. However, the evidence of possible beneficial effects of probiotics, including on UTI incidence in KT patients is missing.

Protocol

All Adult, Caucasian patients treated with kidney transplantation (KT) at SOC Clinica Chirurgica, ASUFC, Udine, Italy, from September 2024, and with an uneventful course during the first postoperative month (POM) will be evaluated for enrollment. Written informed consent to take part in the study will be obtained from each participant after being informed on study design, aims and potential adverse events.

The 132 subjects will be randomly allocated to either the probiotic arm or the placebo arm (control group). Group allocation will be double-blind. A computer random number algorithm (1:1 allocation ratio) will randomize participants, using blocks of four.

In the intervention group, patients will receive two sachets daily of OMNi-BiOTiC® 41167 for 6 months, while the control group will receive an equal amount of similar looking and tasting placebo.

Both study groups will remain on their standard diet and drug regimen during the study period. Adherence to therapy will be measured by sachet count.

The post-transplant clinical surveillance will follow the routine follow-up schedule for KT patients at the Department of Nephrology, ASUFC, Udine, Italy.

At enrollment (POM 1, visit 1) patients will be assessed with routine physical examination, clinical interview, blood exams, tacrolimus dosage and plasma concentration, Torque Teno Virus (TTV) and Acellular Growth Retardation Assay (AGRA) tests, urine tests, urine culture; Nova Food Frequency Questionnaires (NFFQ), Acute Cystitis Symptom Score (ACSS), Gastrointestinal Symptom Rating Scale, Irritable Bowel Syndrome version (GSRS-IBS, AstraZeneca R&D, SE-431 83 Mölndal, Sweden.) and quality of life SF-12 (Hogrefe Verlag, Göttingen, Germany) questionnaires will be administered; clinical data and laboratory data will be collected and saved in dedicated database; urine and stool samples will be collected and stored for microbiota determination; study product will be provided.

BK virus surveillance according to the routine follow-up schedule will be based on viral load measurement in blood and urine samples at POM 1, 3 and 6.

During the treatment period (POM1-POM7, visits 2-15) patients will be assessed with physical examination, routine blood exams, tacrolimus dosage and plasma concentration, urine tests, urine culture; ACSS, GSRS-IBS and SF-12 questionnaires will be administered; clinical data and laboratory data will be collected and saved in dedicated database. Study products will be provided regularly every fourth week.

At the end of the treatment (POM7, visit 16) patients will be assessed with physical examination, routine blood exams, tacrolimus dosage and plasma concentration, TTV and AGRA tests, urine tests, urine culture; NFFQ, ACSS, GSRS-IBS and SF-12 questionnaires will be administered; clinical data and laboratory data will be collected and saved in dedicated database; urine and stool samples will be collected and stored for microbiota determination.

Adverse events and serious adverse events will be evaluated at every visit.

ELIGIBILITY:
Inclusion Criteria:

* willingness and capability to provide written informed consent/assent for the trial;
* ≥18 and <75 years of age on day of signing informed consent;
* patients at 30 days post kidney transplantation with surgically uneventful course during the first postoperative month

Exclusion Criteria:

* pediatric patients (<18 years)
* elderly patients (>75 years)
* combined transplantation recipients
* patients with pre-transplant inflammatory bowel disease or irritable bowel syndrome (according to Roma criteria), previous bowel resection or stoma;
* pre-/probiotic supplementation within 1 month of study commencement or use of other probiotics-containing products during the intervention period;
* any proven gastrointestinal infection or disorder during the first post-transplant month or at the time of study enrollment;
* any surgical complication during the first post-transplant month or at the time of study enrollment;
* evidence of ongoing acute rejection, urinary tract infection or other medical complications at the time of enrollment
* known intolerance or allergy to any of the ingredients in both OMNi-BiOTiC® 41167 and placebo

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infection rates | from postoperative month 1 to postoperative month 7
  UTI will be diagnosed based on seriated urine microbiological cultures. Type of bacteria isolated, bacterial load and antibiogram will be also recorded and confronted
Rates of Urinary tract symptoms | from postoperative month 1 to postoperative month 7
  Urinary tract symptoms will be assessed and diagnosed with seriated ACSS (Acute Cystitis Symptom Score, 0-39; the higher the score, the worse the severity) questionnaires

SECONDARY OUTCOMES:
Rate of biopsy proven acute rejection | from postoperative month 1 to postoperative month 7
  Acute rejection diagnosis will be based on histopathological examination of graft specimen from percutaneous graft biopsy
Immunosuppression therapy | from postoperative month 1 to postoperative month 7
  Immunosuppression therapy will be evaluated with seriated measurements of tacrolimus dosage-to-plasma concentration (TAC-D/C) ratios
Immunosuppression strength | from postoperative month 1 to postoperative month 7
  Immunosuppression strength will be evaluated with seriated plasma AGRA and TTV levels.
Kidney graft function | from postoperative month 1 to postoperative month 7
  Kidney graft function will be assessed with creatinine serum levels
Gut microbiome | at postoperative month 1 and postoperative month 7
  Gut microbiome will be determined by 16S analysis: variation of alpha and beta diversity will be assessed
Bladder microbiome | at postoperative month 1 and postoperative month 7
  Bladder microbiome will be determined by 16S analysis: variation of alpha and beta diversity will be assessed

OTHER OUTCOMES:
Quality of life according to SF-12 questionnaire | from postoperative month 1 to postoperative month 7
  Quality of life will be evaluated with seriated SF-12 (Short form health survey) questionnaires;
Gastrointestinal symptoms according to GSRS-IBS questionnaire | from postoperative month 1 to postoperative month 7
  GI symptoms will be evaluated with seriated GSRS-IBS (The Gastrointestinal Symptom Rating Scale-Irritable Bowel Syndrome) questionnaires
Adverse events | from postoperative month 1 to postoperative month 7
  Incidence of related and unrelated adverse event will be evaluated as a composite outcome based on evidence of abnormal physical examination findings, abnormal laboratory tests results, abnormal imaging examination and/or abnormal microbiological analysis

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Baccarani, MD PhD, Principal Investigator — Department of Medicine, University of Udine; Riccardo Pravisani, MD PhD, Principal Investigator — Department of Medicine, University of Udine; Patrizia Tulissi, MD, Study Director — Azienda Sanitaria Universitaria Friuli Centrale
Locations (1):
- Presidio Ospedaliero Universitario S. Maria della Misericordia, ASUFC, Udine, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winichakoon P, Chaiwarith R, Chattipakorn N, Chattipakorn SC. Impact of gut microbiota on kidney transplantation. Transplant Rev (Orlando). 2022 Jan;36(1):100668. doi: 10.1016/j.trre.2021.100668. Epub 2021 Oct 18. PMID 34688985
- [Background] Liu S, Liu H, Chen L, Liang SS, Shi K, Meng W, Xue J, He Q, Jiang H. Effect of probiotics on the intestinal microbiota of hemodialysis patients: a randomized trial. Eur J Nutr. 2020 Dec;59(8):3755-3766. doi: 10.1007/s00394-020-02207-2. Epub 2020 Feb 28. PMID 32112136
- [Background] Gibson GR, Hutkins R, Sanders ME, Prescott SL, Reimer RA, Salminen SJ, Scott K, Stanton C, Swanson KS, Cani PD, Verbeke K, Reid G. Expert consensus document: The International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of prebiotics. Nat Rev Gastroenterol Hepatol. 2017 Aug;14(8):491-502. doi: 10.1038/nrgastro.2017.75. Epub 2017 Jun 14. PMID 28611480
- [Background] Zaza G, Dalla Gassa A, Felis G, Granata S, Torriani S, Lupo A. Impact of maintenance immunosuppressive therapy on the fecal microbiome of renal transplant recipients: Comparison between an everolimus- and a standard tacrolimus-based regimen. PLoS One. 2017 May 24;12(5):e0178228. doi: 10.1371/journal.pone.0178228. eCollection 2017. PMID 28542523
- [Background] Coussement J, Maggiore U, Manuel O, Scemla A, Lopez-Medrano F, Nagler EV, Aguado JM, Abramowicz D; European Renal Association-European Dialysis Transplant Association (ERA-EDTA) Developing Education Science and Care for Renal Transplantation in European States (DESCARTES) working group and the European Study Group for Infections in Compromised Hosts (E; COLLABORATORS (IN ALPHABETICAL ORDER); European Renal Association-European Dialysis Transplant Association (ERA-EDTA) Developing Education Science and Care for Renal Transplantation in European States (DESCARTES) working group and the European Study Group for Infections in Compromised Hosts (ESGICH) of the European Society of Clinical Microbiology and Infectious Diseases (ESCMID). Diagnosis and management of asymptomatic bacteriuria in kidney transplant recipients: a survey of current practice in Europe. Nephrol Dial Transplant. 2018 Sep 1;33(9):1661-1668. doi: 10.1093/ndt/gfy078. PMID 29635410
- [Background] Eikmans M, Gielis EM, Ledeganck KJ, Yang J, Abramowicz D, Claas FFJ. Non-invasive Biomarkers of Acute Rejection in Kidney Transplantation: Novel Targets and Strategies. Front Med (Lausanne). 2019 Jan 8;5:358. doi: 10.3389/fmed.2018.00358. eCollection 2018. PMID 30671435
- [Background] Garcia-Martinez Y, Borriello M, Capolongo G, Ingrosso D, Perna AF. The Gut Microbiota in Kidney Transplantation: A Target for Personalized Therapy? Biology (Basel). 2023 Jan 20;12(2):163. doi: 10.3390/biology12020163. PMID 36829442
- [Background] Przybycinski J, Drozdzal S, Wilk A, Dziedziejko V, Szumilas K, Pawlik A. The Effect of the Gut Microbiota on Transplanted Kidney Function. Int J Mol Sci. 2023 Jan 9;24(2):1260. doi: 10.3390/ijms24021260. PMID 36674775
- [Background] Strohaeker J, Aschke V, Koenigsrainer A, Nadalin S, Bachmann R. Urinary Tract Infections in Kidney Transplant Recipients-Is There a Need for Antibiotic Stewardship? J Clin Med. 2021 Dec 31;11(1):226. doi: 10.3390/jcm11010226. PMID 35011966
- [Background] Tamargo CL, Kant S. Pathophysiology of Rejection in Kidney Transplantation. J Clin Med. 2023 Jun 19;12(12):4130. doi: 10.3390/jcm12124130. PMID 37373823
- [Background] Ye J, Yao J, He F, Sun J, Zhao Z, Wang Y. Regulation of gut microbiota: a novel pretreatment for complications in patients who have undergone kidney transplantation. Front Cell Infect Microbiol. 2023 Jun 6;13:1169500. doi: 10.3389/fcimb.2023.1169500. eCollection 2023. PMID 37346031